CLINICAL TRIAL: NCT04122664
Title: Prospective Randomized Controlled Study Measuring Posterior Capsular Opacification, Lens Glistenings, Tilt and Decentration, and Visual Outcomes Following Insertion of the RayOne Hydrophobic Lens 800C and the RayOne Hydrophilic Lens 600C.
Brief Title: Posterior Capsular Opacification and Glistenings in Hydrophobic and Hydrophilic Intraocular Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: City, University of London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 265864
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Cataract; Intraocular Lens Opacification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients randomised into one of two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RayOne® Hydrophilic lens 600C (Active Comparator): Patients will be randomly selected to receive the monofocal, acrylic, RayOne® Hydrophilic lens 600C
  Interventions: Device: RayOne® Hydrophilic lens 600C
- RayOne® Hydrophobic lens 800C (Active Comparator): Patients will be randomly selected to receive the monofocal, acrylic, RayOne® Hydrophobic lens 800C
  Interventions: Device: RayOne® Hydrophobic lens 800C

INTERVENTIONS:
Device: RayOne® Hydrophobic lens 800C — Patients will receive a monofocal, aspheric, hydrophobic acrylic intraocular lens: the RayOne® Hydrophobic lens 800C
  Arms: RayOne® Hydrophobic lens 800C
Device: RayOne® Hydrophilic lens 600C — Patients will receive a monofocal aspheric, hydrophilic acrylic intraocular lens: the RayOne® Hydrophilic lens 600C.
  Arms: RayOne® Hydrophilic lens 600C

SUMMARY:
A prospective randomized controlled clinical study to measure posterior capsular opacification, objective measurement of glistenings and intraocular lens tilt and decentration as well as visual outcomes following insertion of a monofocal, aspheric, hydrophobic acrylic intraocular lens: the RayOne® Hydrophobic lens 800C and a monofocal aspheric, hydrophilic acrylic intraocular lens: the RayOne® Hydrophilic lens 600C

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral or bilateral cataracts requiring surgical intervention
2. Age over 18 years
3. Able to understand informed consent and the objectives of the trial
4. Not pregnant, not breast feeding
5. No previous eye surgery
6. Corneal astigmatism less than 1 diopter in both eyes.

Exclusion Criteria:

1. age-related macula degeneration
2. glaucoma
3. previous retinal vascular disorders
4. previous retinal detachment or tear
5. any neuro-ophthalmological condition
6. any inherited retinal disorder or pathology
7. previous strabismus surgery or record of amblyopia
8. previous TIA, CVA or other vaso-occlusive disease
9. already enrolled in another study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2019-10-14 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Posterior Capsular Opacification of Intraocular Lens | 24 months
  Degree of the Posterior Capsular Opacification of Intraocular Lens will be assessed using digital imaging techniques
Intraocular lens glistenings | 24 months
  Degree of the intraocular lens glistenings will be quantified using digital analysis
Intraocular lens tilt and decentration | 24 months

SECONDARY OUTCOMES:
Visual Acuities | 24 months
  Unaided and Best corrected Logmar Visual acuity for distance, and for near vision will be assessed
Forward light scatter and Contrast Sensitivity Measurement | 24 months
  Forward light scatter and Contrast Sensitivity Measurement will be quantified using computerised visual testing
Patient Satisfaction | 24 months
  Validated questionnaires will be used to assess patient satisfaction
Intraoperative and post operative complications | 0 days-24 months

IPD SHARING:
Plan to Share IPD: No